CLINICAL TRIAL: NCT06431347
Title: Prospective Observational Cohort Study of Transplant and Cell Therapy Candidates and Recipients to Assess Social Determinants of Health
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0038; NCI-2024-04536 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-05-22; First posted 2024-05-28 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Transplant and Cell Therapy
Keywords: Social Determinants of Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transplant and Cell Therapy Candidates and Recipients: Participants that agree to take part in this study, the study staff will first verify your demographic information (such as age, sex, race, and so on). Participants will then be asked about social barriers to care, including but not limited to:
  * primary language and confidence speaking English
  * education level
  * employment history
  * health literacy
  * legal history
  * caregiver status and literacy
  Interventions: Behavioral: Social Determinants of Health Questionnaire

INTERVENTIONS:
Behavioral: Social Determinants of Health Questionnaire — Participants will also complete a questionnaire about financial barriers to care within the past year, including income bracket and difficulty affording cost-of-living or medical expenses.

SUMMARY:
To learn more about social and financial factors that may influence outcomes of TCT treatment at MD Anderson.

DETAILED DESCRIPTION:
Primary Objective:

To determine the relationship between participant social determinants of health (SDOH) and outcomes following transplantation and cellular therapy at MDACC.

ELIGIBILITY:
Inclusion Criteria

1. ≥ 18 years of age.
2. Received financial clearance for TCT.

Qualitative study - patients

1. Patient ≥ 18 years of age who is currently cared for at MD Anderson as a TCT candidate/ recipient,
2. The patient reports social and/or financial challenges impacting care delivery.
3. The patient is willing to participate in a semi-structured interview.

Qualitative study - caregivers

1. Caregiver(s) of a patient ≥ 18 years of age who is currently cared for at MD Anderson as a TCT candidate/ recipient.
2. The patient reports social and/or financial challenges impacting care delivery.
3. The patient has referred the caregiver(s) to participate and provided us with permission to contact their caregiver(s).
4. The caregiver(s) is (are) willing to participate in a semi-structured interview.

Exclusion Criteria Patients - Quantitative study 1) Did not receive financial clearance for TCT

Patients - Qualitative study

1) Not impacted by social or financial challenges.

Caregivers (qualitative study)

1. Did not care for a patient impacted by social or financial challenges
2. Were not referred to participate in the study by patient they cared for.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Social Determinants of Health Questionnaire | At 6, 12, 18, and 24 months post Transplant and Cell Therapy

CONTACTS AND LOCATIONS:
Overall Officials: Warren Fingrut, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org